CLINICAL TRIAL: NCT07108699
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Clinical Study to Evaluate the Efficacy and Safety of HSK39004 Dry Powder Inhaler in the Treatment of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Evaluation of the Safety and Efficacy of HSK39004 Dry Powder Inhaler in Chinese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK39004-T1-202
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK39004-0.75mg BID (Experimental)
  Interventions: Drug: HSK39004 Dry Powder Inhaler-0.75mg
- HSK39004-1.5mg BID (Experimental)
  Interventions: Drug: HSK39004 Dry Powder Inhaler-1.5mg
- Placebo control (Experimental)
  Interventions: Drug: HSK39004 Dry Powder Inhaler Simulant

INTERVENTIONS:
Drug: HSK39004 Dry Powder Inhaler-0.75mg — HSK39004 Dry Powder Inhaler: Inhale through the mouth, 0.75mg each time, twice a day
  Arms: HSK39004-0.75mg BID
Drug: HSK39004 Dry Powder Inhaler-1.5mg — HSK39004 Dry Powder Inhaler: Inhale through the mouth, 1.5mg each time, twice a day
  Arms: HSK39004-1.5mg BID
Drug: HSK39004 Dry Powder Inhaler Simulant — HSK39004 Dry Powder Inhaler Simulants, administered via oral inhalation, 1 tablet each time, twice daily
  Arms: Placebo control

SUMMARY:
To evaluate the safety and efficacy of the HSK39004 Dry Powder Inhaler compared with the placebo in the treatment of Chinese patients with COPD.

DETAILED DESCRIPTION:
o evaluate the efficacy, PK characteristics and safety of different doses of HSK39004 Dry Powder Inhaler in patients with COPD under background treatment (single bronchodilator/double bronchodilator, with the combined use of ICS not exceeding 25% of the total enrolled population)

ELIGIBILITY:
Inclusion Criteria:

* 1) During the screening visit (Visit 1), the age range is 40 to 80 years (including the threshold value), and gender is not restricted; 2) The body mass index is within the range of 18 to 30 kg/m2 (including the threshold value); 3) The subjects with chronic obstructive pulmonary disease (COPD) as per the GOLD 2025 diagnostic criteria, and the symptoms before screening were consistent with COPD for at least 1 year [GOLD 2025 standard: the subjects have chronic respiratory symptoms such as shortness of breath, chronic cough or expectoration, and/or have a history of exposure to risk factors, and the pulmonary function test results show: the forced expiratory volume in one second (FEV1) after using bronchodilators / forced vital capacity (FVC) <0.7]; 4) During the screening visit (Visit 1):

  * FEV1/FVC after using bronchodilators is <0.7;
  * 30% of the expected value ≤ FEV1 after using bronchodilators < 80% of the expected value; Note: Using bronchodilators refers to using 400 μg (4 puffs, 100 μg per puff, with an interval of 1 minute between each puff) salbutamol inhalation aerosol for 15 to 30 minutes after use.

    5) At the time of screening, the modified British Medical Research Council (mMRC) dyspnea scale score is ≥ 2; 6) Before screening, at least use bronchodilator drugs for stabilization (single bronchodilator/double bronchodilator, with or without ICS) for ≥ 1 month, and agree to continue using during the study without changing the dosage and type of medication; The prohibited/limited drugs and time intervals before screening are detailed in Chapters 5.9.2 and 5.9.3; 7) During the screening period and treatment period, COPD drugs prohibited by the protocol (except for salbutamol inhalation aerosol as a rescue drug) can be discontinued; 8) Current smokers with a smoking quantity of ≥ 10 packs per year (smoking index (pack years) = daily smoking quantity (packs) × time (years), 1 pack = 20 cigarettes), or former smokers (for example: at least 1 pack per day, for 10 years), or those with a history of exposure to other risk factors.

Exclusion Criteria:

* 1) During the screening visit (Visit 1), the age range is 40 to 80 years (including the threshold value), and gender is not restricted; 2) The body mass index is within the range of 18 to 30 kg/m2 (including the threshold value); 3) The subjects with chronic obstructive pulmonary disease (COPD) as per the GOLD 2025 diagnostic criteria, and the symptoms before screening were consistent with COPD for at least 1 year [GOLD 2025 standard: the subjects have chronic respiratory symptoms such as shortness of breath, chronic cough or expectoration, and/or have a history of risk factor exposure, and the pulmonary function test results show: the forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) after using bronchodilators is less than 0.7]; 4) During the screening visit (Visit 1):

  * FEV1/FVC is less than 0.7 after using bronchodilators;
  * 30% of the expected value ≤ FEV1 < 80% of the expected value after using bronchodilators; Note: Using bronchodilators refers to inhaling 400 μg (4 puffs, 100 μg per puff, with an interval of 1 minute between each puff) salbutamol inhaler for 15 to 30 minutes.

    5) At the time of screening, the modified British Medical Research Council (mMRC) dyspnea scale score is ≥ 2; 6) Before screening, the subjects have been using bronchodilator drugs for stabilization for at least 1 month, and agree to continue using them during the study without changing the dosage and type of medication; The prohibited/limited drugs and time intervals before screening are detailed in Chapters 5.9.2 and 5.9.3; 1) Have a history of life-threatening COPD, including being admitted to the intensive care unit and/or requiring intubation; 2) Have received treatment for COPD acute exacerbation or been hospitalized for pneumonia within 12 weeks before screening; 3) Have had acute (viral or bacterial) upper or lower respiratory tract infections or other infectious diseases requiring antibiotic treatment within 6 weeks before screening; 4) Have other diagnosed respiratory system diseases other than COPD, including but not limited to: α-1 antitrypsin deficiency, asthma, active tuberculosis, lung edema, cystic fibrosis, bronchiectasis, pulmonary nodular disease, or clinically significant pulmonary fibrosis, pulmonary hypertension, interstitial lung disease, bronchiectasis (excluding asymptomatic local bronchial dilation); 5) Have a history of or currently have severe cardiovascular diseases, including but not limited to:
  * Screening period NYHA cardiac function grade III/IV (according to the NYHA cardiac function grading standard, see Appendix 1);
  * Had acute myocardial infarction, unstable angina pectoris/acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass grafting within 6 months before screening;
  * Structural heart disease, such as hypertrophic cardiomyopathy, moderate to severe valvular disease;
  * Had severe arrhythmia within 3 months before screening, such as: atrial fibrillation with a ventricular rate > 120 bpm, ventricular tachycardia, bradycardia (ventricular rate < 45 bpm), second-degree II or above atrioventricular conduction block (excluding those with implanted pacemaker or defibrillator), male QTcF > 450 ms or female QTcF > 470 ms;
  * Subjects with poor blood pressure control (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg at the screening visit); 6) Have type I diabetes or poorly controlled type II diabetes (fasting blood glucose ≥ 10 mmol/L at screening); 7) Have cancer (in situ cancer that has been cured for more than 5 years, skin squamous cell carcinoma and basal cell carcinoma, etc., except for subjects with suspected malignant tumors or undetermined tumors); 8) Combine other severe unstable kidney, nervous system, endocrine diseases, thyroid diseases, urinary system, ophthalmic diseases, immune system, mental system, gastrointestinal, liver or blood system disease/abnormal history, as determined by the investigator, participation in this study may pose risks to the subjects or affect the analysis of research results; 9) During the screening period (visit 1), the investigator determines that the laboratory tests of the subjects show clinically significant abnormalities that may pose risks to the subjects, including but not limited to the following situations:

    1. The glomerular filtration rate (eGFR) calculated using the CKD-EPI formula is less than 60 mL/min/1.73m2;
    2. Liver function: Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) are more than 2.5 times the upper limit of the normal value; Total bilirubin (TBIL) is more than 1.5 times the upper limit of the normal value.

       10) Lactose/milk protein (dairy products) intolerance, allergy to HSK39004 inhalation powder or salbutamol or any known components in the administration system; 11) Before the pulmonary function test during the screening (visit 1), any prohibited drugs in the protocol were used (see Table 4 and Table 5 of the prohibited drug list in Section 5.9.3); 12) Within 12 months before screening, received lobectomy or lung volume reduction surgery; 13) Had major surgery (requiring general anesthesia) within 6 weeks before screening, not fully recovered at the time of screening, or planned to undergo surgery before the end of the study; 14) Patients determined by the investigator to require oxygen therapy; 15) Have clinically significant apnea that requires the use of a continuous airway positive pressure ventilation (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The ΔFEV1 AUC0-12h after the 4th week administration (the area under the curve representing the change in FEV1 from baseline to 12 hours after administration) | Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China